CLINICAL TRIAL: NCT04922502
Title: Parent-based Treatment for Youth With Anxiety and Obsessive-compulsive Disorder: Comparison of Therapist-Led and Therapist Assisted Approaches
Brief Title: Parent-based Treatment for Youth With Anxiety and Obsessive-compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-49809
Record Dates: First submitted 2021-05-25; First posted 2021-06-10 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Obsessive-Compulsive Disorder in Children; Social Anxiety Disorder of Childhood; Obsessive-Compulsive Disorder in Adolescence; Separation Anxiety; Generalized Anxiety Disorder; Panic Disorder; Panic Attacks; Panic With Agoraphobia
Keywords: obsessive-compulsive disorder; children; cognitive behavioral therapy; anxiety
MeSH Terms: conditions — Anxiety, Separation; Generalized Anxiety Disorder; Panic Disorder; Obsessive-Compulsive Disorder; Anxiety Disorders | interventions — Bibliotherapy

STUDY DESIGN:
Intervention Model Description: Randomized assignment to one of two conditions
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard SPACE (Active Comparator): 12 one hour parent sessions over 12 weeks in which the therapist guides the parent to target anxious behaviors and support adaptive child behaviors.
  Interventions: Behavioral: Standard SPACE
- Bibliotherapy, low therapist contact SPACE (Active Comparator): 4 one hour parent sessions over 12 weeks in which the therapist supports the parent in understanding and implementing content reviewed in the book "Breaking Free of Child Anxiety and OCD".
  Interventions: Behavioral: Bibliotherapy, low therapist contact SPACE

INTERVENTIONS:
Behavioral: Standard SPACE — 12 one hour parent sessions over 12 weeks in which the therapist guides the parent to target anxious behaviors and support adaptive child behaviors.
  Arms: Standard SPACE
Behavioral: Bibliotherapy, low therapist contact SPACE — 4 one hour parent sessions over 12 weeks in which the therapist supports the parent in understanding and implementing content reviewed in the book "Breaking Free of Child Anxiety and OCD".
  Arms: Bibliotherapy, low therapist contact SPACE

SUMMARY:
Anxiety and obsessive-compulsive disorders are the most common mental health disorders in childhood and adolescence. A parenting intervention for youth with anxiety, called Supportive Parenting of Anxious Childhood Emotions ("SPACE"), has been recently developed to help target anxiety in children. In this intervention, therapists meet individually with parents to help them reduce anxiety behaviors in their children and support adaptive behaviors in their children. The purpose for the proposed study is to demonstrate the treatment efficacy of SPACE compared to a low-contact, therapist-supported bibliotherapy version of this intervention.

DETAILED DESCRIPTION:
Anxiety and obsessive-compulsive disorders are the most common mental health disorders in childhood and adolescence. Parental accommodation of their children's avoidance, escape, safety behaviors are a set of parenting behaviors that have been most strongly associated with child anxiety and obsessive-compulsive disorder. Developing and testing parent-led interventions that target accommodation and parenting styles associated with anxiety has the potential to improve treatment outcomes and reach families who may not otherwise access care (for example, for youth who refuse to attend therapy). A parenting intervention for youth with anxiety has been recently developed to address these goals called Supportive Parenting of Anxious Childhood Emotions ("SPACE"). In this intervention, therapists meet individually with parents to help them reduce accommodation and support adaptive behaviors in their children. SPACE was recently shown to be non-inferior to individual cognitive-behavioral therapy with 88% of youth being classified as responders to SPACE. The purpose for the proposed study is to demonstrate the treatment efficacy of SPACE compared to a low-contact, therapist-supported bibliotherapy version of this intervention, providing efficacy evidence for SPACE as delivered by an independent investigatory group.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 7 to 17 at enrollment
* The child has clinically significant symptoms of anxiety and/or OCD, as indicated by a score of 12 or higher on the Pediatric Anxiety Rating Scale (PARS).
* The child is appropriate for anxiety-focused treatment (e.g., anxiety is the primary problem as diagnosed using the Anxiety Disorders Interview Schedule (ADIS), and if secondary psychopathology is present it will not interfere with treatment).
* One parent/guardian is able and willing to participate in assessment and treatment (e.g., has sufficient English fluency, the decisional capacity to participate, and can commit to treatment duration).
* The participating parent/guardian lives with their child at least 50% of the time.
* Both parent and child are able to read and understand English.
* The child is able to communicate verbally.
* Participants must reside in Texas and parents must be in the state of Texas when taking calls.

Exclusion Criteria:

* the child has a diagnosis of child lifetime bipolar disorder, drug of alcohol abuse, intellectual or developmental disability, psychotic disorder, or conduct disorder.
* the child has severe, current suicidal/homicidal ideation and/or self-injury requiring medical intervention (referrals will be made for appropriate clinical intervention).
* the child is receiving concurrent evidence-based psychotherapy for anxiety, involving exposure therapy in at least 50% of sessions.
* the child has initiated or changed dosage of psychotropic medications within 4 weeks before study enrollment OR stimulant or benzodiazepine medications within 2 weeks before study enrollment. If appropriate, the child may be enrolled in the study once medication dosage has stabilized (i.e., 4 weeks for psychotropic medication or 2 weeks for stimulant/benzodiazepine medication).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Storch EA, Guzick AG, Ayton DM, Palo AD, Kook M, Candelari AE, Maye CE, McNeel M, Trent ES, Garcia JL, Onyeka OC, Rast CE, Shimshoni Y, Lebowitz ER, Goodman WK. Randomized trial comparing standard versus light intensity parent training for anxious youth. Behav Res Ther. 2024 Feb;173:104451. doi: 10.1016/j.brat.2023.104451. Epub 2023 Dec 17. PMID 38154287

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment numbers reflect both parent and child of the parent-child dyads.
Period: Overall Study
Arm/Group | Standard SPACE | Bibliotherapy, Low Therapist Contact SPACE
Started (No cross-over between Bibliotherapy, Low Therapist Contact SPACE to Standard SPACE occurred.) | 66 (Sample reflects parent-child dyads including 33 parents and 33 children.) | 70 (Sample reflects parent-child dyads including 35 parents and 35 children.)
Completed | 60 (Sample reflects parent-child dyads including 30 parents and 30 children.) | 62 (Sample reflects parent-child dyads including 31 parents and 31 children.)
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were not collected for Parents and only reflect the Child.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard SPACE | Bibliotherapy, Low Therapist Contact SPACE | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 35 | 68
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.6) | 10.2 (2.8) | 10.2 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 21 | 21 | 42
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 35 | 68
Clinical Global Impressions Scale-Severity [Mean (Standard Deviation); unit: units on a scale] — 7 point scale ranging from 0 (no illness) to 6 (most severe patient seen)
  units on a scale | 3.48 (.67) | 3.54 (.82) | 3.51 (.74)
Pediatric Anxiety Rating Scale-Revised [Mean (Standard Deviation); unit: units on a scale] — The Pediatric Anxiety Rating Scale-Revised (PARS) includes a 59-item symptom checklist and 7-item severity scale with parent and clinician-rated scores with range from 0 to 35. Higher scores indicate higher symptom severity.
  units on a scale | 17.63 (2.67) | 16.51 (4.14) | 17.06 (3.52)

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anxiety Rating Scale
Description: Clinician-rated child anxiety severity throughout the past week. Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 35.
Time Frame: Baseline (before treatment), post-treatment assessment (on average 12 weeks), one month follow up; Baseline scores reported.
Population: Three participants did not complete the standard SPACE intervention, and 4 participants did not complete the low-therapist contact SPACE intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard SPACE | Bibliotherapy, Low Therapist Contact SPACE
Number analyzed (Participants) | 30 | 31
score on a scale | 10.86 (4.80) | 10.96 (6.08)

2. Secondary Outcome: Anxiety Disorders Interview Schedule (ADIS-IV) With Clinical Severity Ratings
Description: Clinician-rated diagnostic interview that includes current anxiety disorders, depression, obsessive-compulsive disorder, and related disorders. Each diagnostic category is coded as present or absent based on symptom criteria and clinical severity ratings (CSRs), which indicate the level of clinical interference. CSRs are scored on a 0-8 scale (0 = not at all; 8 = very, very much). CSRs of 4 or above indicate the clinical levels.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Clinical Global Impression-Severity
Description: Clinician-rated child psychopathology severity rating. A single item is scored 0-6 (0= no illness; 6= extremely severe symptoms).
Time Frame: as for outcome 1
Population: three participants did not complete the standard SPACE intervention and 4 participants did not complete the low-therapist contact SPACE intervention. Data for baseline scores reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard SPACE | Bibliotherapy, Low Therapist Contact SPACE
Number analyzed (Participants) | 30 | 31
score on a scale | 2.42 (0.89) | 2.52 (0.93)

ADVERSE EVENTS:
Time Frame: Participants were assessed up to 16 weeks. Non-responders to bibliotherapy had the option to participate in standard SPACE, and were possibly followed for an additional 8 weeks (for a total of 24 weeks). Adverse event data were collected for child participants only and were collected for the duration of a participant's involvement in the study.
Description: The definition of an adverse event does not differ from that used on clinicaltrials.gov
Arm/Group | Standard SPACE | Bibliotherapy, Low Therapist Contact SPACE
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 0/33 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT04922502/Prot_SAP_ICF_000.pdf